CLINICAL TRIAL: NCT04673032
Title: Radiofrequency (RF) Ablation Prospective Outcomes Study
Acronym: RAPID
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: A4087
Record Dates: First submitted 2020-12-12; First posted 2020-12-17 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Pain, Chronic
Keywords: Radiofrequency (RF)
MeSH Terms: conditions — Chronic Pain | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Boston Scientific Radiofrequency Ablation Systems: Subjects with pain treated with a commercially approved Boston Scientific RF system
  Interventions: Device: Radiofrequency Ablation

INTERVENTIONS:
Device: Radiofrequency Ablation — Radiofrequency Ablation for treatment of chronic pain

SUMMARY:
The objective of this study is to compile real-world outcomes of Boston Scientific commercially approved radiofrequency (RF) ablation systems in the treatment of patients diagnosed with pain

ELIGIBILITY:
Key Inclusion Criteria:

* Study candidate is scheduled to be treated with a commercially approved Boston Scientific RF system for pain per local Directions for Use (DFU)
* Signed a valid, IRB/EC/REB-approved informed consent form

Key Exclusion Criteria:

* Meets any contraindications per locally applicable Directions for Use (DFU)
* Currently diagnosed with cognitive impairment, or exhibits any characteristic, that would limit study candidate's ability to assess pain relief or to complete study assessments

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Chronic Pain
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Patient Global Impression of Change (PGIC) | 12-months post-procedure
  Using the Patient Global Impression of Change (PGIC) Scale, subjects will rate themselves as: very much improved; much improved; minimally improved; no change; minimally worse; much worse; or very much worse compared with Baseline

OTHER OUTCOMES:
Responder rate | 3-months post-procedure
  Proportion of subjects with a 30 percent or greater reduction from Baseline in targeted pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, M.S., Study Director — Boston Scientific Corporation
Locations (15):
- United States (11):
  - Elite Pain and Spine Institute, Mesa, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - The Spine Wellness Center in Westport, Westport, Connecticut
  - Shepherd Center, Atlanta, Georgia
  - Quincy Medical Group, Quincy, Illinois
  - Twin Cities Pain Clinic and Surgery Center, Edina, Minnesota
  - Carolinas Research Institute, Huntersville, North Carolina
  - UC Health Pain Medicine, Cincinnati, Ohio
  - Premier Pain Treatment Institute, Loveland, Ohio
  - Toledo Clinic, Toledo, Ohio
  - Pain Diagnostics and Interventional Care, Sewickley, Pennsylvania
- Belgium (2):
  - ZNA Hoge Beuken, Antwerp
  - St. Jan, Bruges
- Mater Olbia Hospital, Olbia, Italy
- St. Anna Hospital, Geldrop, Netherlands

REFERENCES:
- [Derived] Provenzano DA, Holt B, Danko M, Atallah J, Iqbal M, Shah B, Singh A, Sachdeva H, Donck EV, Liebrand B, Shaw E, Haas S, Sekhar R, Pan A, Halperin DS, Goldberg E. Assessment of real-world, prospective outcomes in patients treated with cervical radiofrequency ablation for chronic pain (RAPID). Interv Pain Med. 2025 Aug 23;4(3):100623. doi: 10.1016/j.inpm.2025.100623. eCollection 2025 Sep. PMID 40896553
- [Derived] Provenzano DA, Holt B, Danko M, Atallah J, Iqbal M, Shah B, Singh A, Sachdeva H, Donck EV, Shaw E, Haas S, Sekhar R, Pan A, Halperin DS, Goldberg E. Assessment of real-world, prospective outcomes in patients treated with lumbar radiofrequency ablation for chronic pain (RAPID). Interv Pain Med. 2025 Apr 24;4(2):100576. doi: 10.1016/j.inpm.2025.100576. eCollection 2025 Jun. PMID 40342788